CLINICAL TRIAL: NCT05162755
Title: A Phase 1a/1b, Open-label, Multicenter Trial Investigating the Safety, Tolerability, and Preliminary Anti-neoplastic Activity of S095029 (Anti-NKG2A) as Monotherapy and in Combination With Sym021 (Anti-PD-1) in Patients With Advanced Solid Tumor Malignancies Followed by an Expansion Part With Triplet Combinations of S095029 and Sym021 and an Anti-HER2 mAb or Anti-EGFR mAbs (Futuximab/Modotuximab) in Patients With Metastatic Gastric or Colorectal Cancers
Brief Title: S095029 as Monotherapy and in Combination With Sym021 in Patients With Advanced Solid Tumor Malignancies Followed by an Expansion Part With Triple Combinations in Patients With Metastatic Gastric or Colorectal Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95029-001
Record Dates: First submitted 2021-10-14; First posted 2021-12-17 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
Keywords: Adults; Advanced solid tumors; Sym21; Futuximab/modotuximab; Triplet combination; Anti-EGFR; Anti-HER2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation 1a: S95029 (Experimental)
  Interventions: Drug: S095029
- Dose escalation 1b: S95029 and Sym021 (Experimental)
  Interventions: Drug: S95029 and Sym021

INTERVENTIONS:
Drug: S095029 — S095029 will be administered via IV infusion every 2 weeks. Once the DLT evaluations period at the second dose level is completed and it is deemed as safe, the dose escalation part 1b will be initiated.
  Arms: Dose escalation 1a: S95029
Drug: S95029 and Sym021 — Sym021 will be administered at a fixed dose of 200mg. S095029 will be administered via IV infusion every 2 weeks. Once the RP2D dose of S95029 in combination with Sym21 is defined, dose expansion will begin.
  Arms: Dose escalation 1b: S95029 and Sym021

SUMMARY:
The purpose of the study is to investigate the safety, tolerability, and preliminary anti-neoplastic activity of S095029 alone and in combination with Sym021 in patients with advanced solid tumor malignancies followed by an expansion phase of triple combinations.

*The study sponsor has made the decision not to move forward to the expansion part of the study due to strategic considerations, unrelated to any safety issues or concerns. The study will be stopped after completion of dose escalation parts 1a and 1b of the study.

ELIGIBILITY:
Dose escalation part:

Inclusion Criteria:

* Histologically or cytologically confirmed unresectable, locally advanced or metastatic solid tumor malignancies
* Patients with a malignancy not amenable to surgical intervention
* Patients with measurable disease and progression radiologically assessed
* Patients with disease progression after treatment with available standard of care therapies that are known to confer clinical benefit or who are intolerant to treatment.
* Patients with available archived tumor biopsy specimens or agree to mandatory biopsy
* Estimated life expectancy ≥ 12 weeks
* Adequate haematological function
* Adequate renal function
* Adequate hepatic function

Exclusion Criteria:

* Pregnant and lactating women
* Major surgery within 4 weeks prior to the first IMP administration or not recovered from the surgery
* Patients with serious/active/uncontrolled infection or infection requiring parenteral antibiotics, within 2 weeks prior to first IMP administration
* Active Hepatitis B Virus infection
* Carriers of HIV antibodies
* Patients with active thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 4 weeks prior to first IMP administration
* History of organ transplantation
* History of gastrointestinal perforation, or intra-abdominal abscess within 28 days of inclusion
* History of cirrhosis
* History of pulmonary fibrosis or relevant uncontrolled chronic pulmonary condition
* Treatment with systemic immunosuppressive therapy
* Active autoimmune disease
* Administration of a live vaccine within 28 days prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) (Dose escalation part) | Through study completion, up to 2 years
  Incidence, severity, and relationship of AEs
Incidence of dose limiting toxicities (DLTs) (Dose escalation part) | At the end of Cycle 1 (each cycle is 28 days)
  DLTs observed during a 28-day period

SECONDARY OUTCOMES:
Objective Response Rate | Through study completion, up to 2 years
Clinical Benefit Rate (CBR) | Through study completion, up to 2 years
  Assessment based on complete response, partial response and stable disease ≥ 6 months
Duration of response (DOR) | Through study completion, up to 2 years
Progression Free Survival (PFS) | Through study completion, up to 2 years
Overall Survival (OS) | Through study completion, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Lakhani MD, MD, PhD, Principal Investigator — Director of Clinical Research START Midwest
Locations (5):
- United States (4):
  - START Midwest, Grand Rapids, Michigan
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The START Center for Cancer Care, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/